CLINICAL TRIAL: NCT02777528
Title: Evaluation of the GORE® TAG® Thoracic Branch Endoprosthesis (TBE Device) in the Treatment of Lesions of the Aortic Arch and Descending Thoracic Aorta, Zone 0/1
Brief Title: Evaluation of the GORE® TBE Device in the Treatment of Lesions of the Aortic Arch and Descending Thoracic Aorta, Zone 0/1
Acronym: SSB 11-02
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSB 11-02 Pivotal (Zone 0/1)
Record Dates: First submitted 2016-05-12; First posted 2016-05-19 (Estimated); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Aortic Aneurysm, Thoracic; Aorta, Lesion
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Zone 0/1 Aortic aneurysm (Other): Zone 0/1 Aortic aneurysm
  Interventions: Device: GORE® TAG® Thoracic Branch Endoprosthesis; Procedure: Revascularization Procedure
- Zone 0/1 Non-aneurysm aortic lesions (Other): Includes dissection and other isolated lesion types
  Interventions: Device: GORE® TAG® Thoracic Branch Endoprosthesis; Procedure: Revascularization Procedure

INTERVENTIONS:
Device: GORE® TAG® Thoracic Branch Endoprosthesis — Endovascular repair with the TBE Device
Procedure: Revascularization Procedure — Revascularization procedure of the great vessel

SUMMARY:
The objective of this study is to determine whether the GORE® TAG® Thoracic Branch Endoprosthesis is safe and effective in treating lesions of the aortic arch and descending thoracic aorta.

DETAILED DESCRIPTION:
For Zone 0/1, there are two arms (Aneurysm arm, Non-aneurysm arm) and three cohorts, described as follows: Zone 0/1 Aneurysm, Zone 0/1 Dissection, and Zone 0/1 Other Isolated Lesion. The Zone 0/1 Aneurysm cohort was the only cohort analyzed with a hypothesis test, however data was collected similarly for all cohorts and for continued access Subjects. Zone 0/1 Subjects enrolled for analysis were from the United States and Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of thoracic aortic pathology deemed to warrant surgical repair which requires proximal graft placement in Zone 0-2.
2. Age ≥18 years at time of informed consent signature
3. Subject is capable of complying with protocol requirements, including follow-up
4. Informed Consent Form (ICF) is signed by Subject or legal representative
5. Must have appropriate proximal aortic landing zone.
6. Must have appropriate target branch vessel landing zone.
7. For patients with aneurysm/isolated lesion, must have appropriate distal aortic landing zone.
8. Native aortic valve (Zone 0/1 subjects only)
9. Subject is considered a high risk candidate for conventional open surgical repair at the discretion of the Investigator (Zone 0/1 subjects only)

Exclusion Criteria:

1. Concomitant disease of the ascending aorta or aneurysm of the abdominal aorta requiring repair
2. Previous endovascular repair of the ascending aorta
3. Previous endovascular repair of the DTA with a non-Gore device
4. Surgery within 30 days prior to enrollment, with the exception of surgery for Ascending Aortic Dissection and/or placement of vascular conduit for access.
5. Infected aorta
6. Life expectancy <2 years
7. Myocardial infarction within 6 weeks prior to treatment
8. Stroke within 6 weeks prior to treatment, stroke defined as rapidly developing clinical signs of focal (or global) disturbance of cerebral function, lasting more than 24 hours or leading to death, with no apparent cause other than that of vascular origin.
9. Patient has a systemic infection and may be at increased risk of endovascular graft infection
10. Pregnant female at time of informed consent signature
11. Degenerative connective tissue disease, e.g. Marfan's or Ehler-Danlos Syndrome
12. Participation in another drug or medical device study within one year of study enrollment
13. Known history of drug abuse within one year of treatment
14. Presence of protruding and/or irregular thrombus and/or atheroma in the aortic arch or ascending aorta
15. Tortuous or stenotic iliac and/or femoral arteries preventing introducer sheath insertion and the inability to use a conduit for vascular access
16. Planned coverage of celiac artery
17. Patient has known sensitivities or allergies to the device materials
18. Patient has known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment
19. Previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or known hypersensitivity to heparin
20. Patient with a history of a hypercoagulability disorder and/or hypercoagulability state
21. Diameter taper outside of the device sizing range between proximal and distal landing zones of aorta and the inability to use additional devices of different diameters to compensate for the taper
22. Mycotic aneurysm
23. Persistent refractory shock (systolic blood pressure <90 mm Hg)
24. Patient has body habitus or other medical condition which prevents adequate visualization of the aorta
25. Renal failure defined as patients with an estimated Glomerular Filtration Rate (eGFR) <30 or currently requiring dialysis
26. Patient at high risk of neurological event, e.g. stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-08; Primary Completion 2024-03 (Actual); Study Completion 2028-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dake, MD, Principal Investigator — Stanford University; Himanshu Patel, MD, Principal Investigator — University of Michigan
Locations (39):
- United States (34):
  - Keck Medical Center of USC, Los Angeles, California
  - Cedar-Sinai Medical Center, Los Angeles, California
  - Leland Stanford Junior University, Stanford, California
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida-Gainesville, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwesten University, Chicago, Illinois
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - University of Baltimore Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington Univeristy School of Medicine - St Louis, St Louis, Missouri
  - Dartmouth-Hitchock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Research Foundation SUNY Buffalo, Buffalo, New York
  - Carolinas HealthCare Systems, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Cardiovascular Surgery Clinic, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Baylor College of Medicine - Houston, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann, Houston, Texas
  - Heart Hospital at Baylor Plano, Plano, Texas
  - Sentara Medical Group, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin System, Madison, Wisconsin
- Japan (5):
  - Nagoya University Hospital, Aichi
  - Morinomiya Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Oita University Hospital, Ōita
  - Jikei Medical University Hospital, Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study enrolled participants into 2 Zones (7 total cohorts) and results are reported by zone. This record (NCT02777528) contains the results for the 3 cohorts of Zone 0/1 (Zone 0/1 Aneurysm Cohort, Zone 0/1 Dissection Cohort, Zone 0/1 Other Isolated Lesion Cohort). Results for the 4 cohorts of Zone 2 (Zone 2 Aneurysm Cohort, Zone 2 Dissection Cohort, Zone 2 Other Lesions Cohort, Zone 2 Traumatic Transection Cohort) are reported in a separate record (NCT02777593).
Groups:
- Zone 0/1 Aneurysm Cohort: Aneurysm arm, hypothesis-driven cohort
- Zone 0/1 Dissection Cohort: Non-aneurysm arm, dissection cohort
- Zone 0/1 Other Isolated Lesion Cohort: Non-aneurysm arm, other isolated lesion cohort
Period: Overall Study
Arm/Group | Zone 0/1 Aneurysm Cohort | Zone 0/1 Dissection Cohort | Zone 0/1 Other Isolated Lesion Cohort
Started | 52 | 24 | 3
Analysis Population (Two participants are excluded from results analysis as pre-specified due to treatment with 49/53 mm device no longer supported by the protocol) | 50 | 24 | 3
Completed | 6 | 4 | 0
Not Completed | 46 | 20 | 3
Not completed — Still in study | 24 | 10 | 1
Not completed — Study Device Explanted | 1 | 0 | 0
Not completed — Death | 14 | 7 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Discontinued due to Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Two Zone 0/1 Aneurysm participants that are counted in the Participant Flow section above are excluded from this analysis, as pre-specified, due to treatment with 49/53 mm device no longer supported by the protocol. As described in the Participant Flow Section, the study reports results in 2 separate records. Zone 2 cohorts are reported in record NCT02777593.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zone 0/1 Aneurysm Cohort | Zone 0/1 Dissection Cohort | Zone 0/1 Other Isolated Lesion Cohort | Total
Number analyzed (Participants) | 50 | 24 | 3 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.3 (8.56) | 63.0 (11.31) | 73.7 (9.02) | 70.8 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 7 | 1 | 26
  Male | 32 | 17 | 2 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 4
  Not Hispanic or Latino | 47 | 23 | 3 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27 | 13 | 3 | 43
  Black or African American | 6 | 6 | 0 | 12
  Asian | 16 | 2 | 0 | 18
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Hawaiian or Pacific Islander | 1 | 1 | 0 | 2
  Other | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 40 | 23 | 3 | 66
  Japan | 10 | 1 | 0 | 11
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Site was queried and the weight for one Zone 0/1 Aneurysm Subject is unavailable.
  kg/m^2
    number analyzed (Participants) | 49 | 24 | 3 | 76
    (all) | 27.3 (5.94) | 29.9 (4.44) | 23.4 (2.01) | 27.9 (5.57)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Primary Endpoint Success Through 1 Month for Zone 0/1
Description: Primary Endpoint was composite of the following events from the time of enrollment through one month following the endovascular procedure (through day 59 unless otherwise specified): initiation of the index endovascular procedure following the debranching procedure, device technical success for the index endovascular procedure and absence of aortic rupture, lesion related mortality, disabling stroke, permanent paraplegia, permanent paraparesis, new onset renal failure requiring permanent dialysis, additional unanticipated post-procedural surgical or interventional procedure related to the device, procedure, or withdrawal of the delivery system. Limited to 30 days: disabling stroke, permanent paraplegia, permanent paraparesis, new onset renal failure requiring permanent dialysis.
Time Frame: 1 month
Population: Two Zone 0/1 Aneurysm participants that are counted in the Participant Flow section above are excluded from this analysis, as pre-specified due to treatment with 49/53 mm devices no longer supported by the protocol.
  Primary Endpoint composite denominator was restricted to number of participants either with a primary endpoint event or imaging performed in the 1 Month window.
Measure: Number; unit: proportion of participants
Arm/Group | Zone 0/1 Aneurysm Cohort | Zone 0/1 Dissection Cohort | Zone 0/1 Other Isolated Lesion Cohort
Number analyzed (Participants) | 47 | 22 | 3
proportion of participants | 0.745 | 0.818 | 1.0
Statistical Analysis 1: Comparison: Zone 0/1 Aneurysm Cohort; Primary endpoint success was defined as the proportion of analysis-eligible participants without a primary endpoint event and with 1-Month imaging performed. Results were tested against a performance goal (PG) of 0.60 (i.e. 60%), derived from outcomes from a systematic review of hybrid TEVAR repair literature. Additionally, using a one-sided alpha of 0.05 and Exact Test, minimum power of 80%, the sample needed was 50 patients; Test type: Other — Performance goal tested using Exact method calculation to estimate the 95% one-sided lower confidence level (95% LCL) on the proportion of participants with primary endpoint success. If the 95% LCL exceeded 0.60, then the null hypothesis was to be rejected and the PG was met; 95% Exact Lower Confidence Limit = 0.745

2. Primary Outcome: Proportion of Participants With Primary Endpoint Success Through 12 Months for Zone 0/1
Description: Primary Endpoint was composite of the following events from the time of enrollment through twelve months following the endovascular procedure: initiation of the index endovascular procedure following the debranching procedure, device technical success for the index endovascular procedure and absence of aortic rupture, lesion related mortality, disabling stroke, permanent paraplegia, permanent paraparesis, new onset renal failure requiring permanent dialysis, additional unanticipated post-procedural surgical or interventional procedure related to the device, procedure, or withdrawal of the delivery system. Limited to 30 days: disabling stroke, permanent paraplegia, permanent paraparesis, new onset renal failure requiring permanent dialysis.
Time Frame: 12 months
Population: Two Zone 0/1 Aneurysm participants that are counted in the Participant Flow section above are excluded from this analysis, as pre-specified, due to treatment with 49/53 devices no longer supported by the protocol.
  Primary Endpoint composite denominator was restricted to number of participants either with a primary endpoint event or imaging performed in the 12 Month window.
Measure: Number; unit: proportion of participants
Arm/Group | Zone 0/1 Aneurysm Cohort | Zone 0/1 Dissection Cohort | Zone 0/1 Other Isolated Lesion Cohort
Number analyzed (Participants) | 44 | 24 | 2
proportion of participants | 0.727 | 0.750 | 1.0

ADVERSE EVENTS:
Time Frame: Adverse events collected for 60 Months, rates shown are through 12-months follow-up, follow-up is ongoing for participants who have not completed the study.
Description: The two excluded Zone 0/1 Aneurysm participants, due to treatment with 49/53 mm device no longer supported by the protocol, have been included in this Adverse Events section.
  Collection starting at revascularization procedure. Adverse event data collection is still ongoing and will be updated upon study completion.
  As described in the Participant Flow Section, the study reports results in 2 separate records. Zone 2 cohorts are reported in record NCT02777593.
Arm/Group | Zone 0/1 Aneurysm Cohort | Zone 0/1 Dissection Cohort | Zone 0/1 Other Isolated Lesion Cohort
All-Cause Mortality (participants affected / at risk) | 14/52 | 7/24 | 1/3
Serious Adverse Events (participants affected / at risk) | 43/52 | 19/24 | 1/3
Other Adverse Events (participants affected / at risk) | 40/52 | 21/24 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zone 0/1 Aneurysm Cohort (N=52) | Zone 0/1 Dissection Cohort (N=24) | Zone 0/1 Other Isolated Lesion Cohort (N=3)
Acute blood loss anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia aggravated (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute systolic heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic regurgitation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Asystole (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Complete heart block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Congestive cardiac failure aggravated (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Pericardial effusion malignant (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Systolic heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Right cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision loss (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Alcoholic gastritis, without mention of hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aortoenteric fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bleeding gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
GI bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mesenteric ischemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal hematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Puncture site bleeding (General disorders) | 1 (1) | 0 (0) | 0 (0)
Stent-graft endoleak type IA (General disorders) | 0 (0) | 1 (1) | 0 (0)
Stent-graft endoleak type IB (General disorders) | 4 (4) | 0 (0) | 0 (0)
Stent-graft endoleak type II (General disorders) | 2 (2) | 0 (0) | 0 (0)
Stent-graft endoleak type IIIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Unknown cause of death (General disorders) | 2 (2) | 2 (2) | 1 (1)
Alcoholic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bilateral pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diarrhea, Clostridium difficile (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gram-positive bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hospital acquired pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective aortitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Inguinal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Klebsiella septicemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nosocomial pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Obstructive pneumonia (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Periapical dental abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (6) | 0 (0) | 0 (0)
Pneumonia aggravated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Vascular graft infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vascular stent graft infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Alcohol intoxication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bladder injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bypass graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bypass graft stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral artery pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fracture of one or more phalanges of hand, open (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incision site hematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Intertrochanteric femoral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intraoperative bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intraoperative venous injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post spinal headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural hematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Tongue laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Degenerative arthritis peripheral joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Knee arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis knees (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid artery dissection (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarct (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischemic stroke (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paralysis vocal cord (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter breakage (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure aggravated (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal hemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Uremia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary bladder hematoma (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0)
Acute on chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bilateral pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercapnic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Increased shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Blood loss of (NOS) (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Blue toe syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis leg (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Descending thoracic aorta rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Descending thoracic aortic aneurysm enlargement (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Dissecting aneurysm of aorta (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Femoral artery dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Hypovolemic shock (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Iliac artery dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Iliac artery rupture (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Leg ischemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Low blood pressure (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zone 0/1 Aneurysm Cohort (N=52) | Zone 0/1 Dissection Cohort (N=24) | Zone 0/1 Other Isolated Lesion Cohort (N=3)
Acute post hemorrhagic anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (3) | 0 (0)
Acute pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (6) | 2 (3) | 0 (0)
Stent-graft endoleak (General disorders) | 2 (2) | 2 (2) | 0 (0)
Stent-graft endoleak type II (General disorders) | 9 (9) | 2 (2) | 0 (0)
Weakness generalized (General disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous graft site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 6 (6) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (8) | 1 (1) | 0 (0)
Appetite lost (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 0 (0) | 0 (0)
Hoarseness of voice (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascending aortic aneurysm enlargement (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Groin hematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 7 (8) | 2 (2) | 0 (0)
Iliac artery dissection (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT02777528/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT02777528/SAP_001.pdf